CLINICAL TRIAL: NCT00137371
Title: Efficacy and Safety of 2 Low-Dose Regimens of Conjugated Estrogen Cream Administered Vaginally in Postmenopausal Women With Atrophic Vaginitis
Brief Title: Study Evaluating Conjugated Estrogen Cream for Atrophic Vaginitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0713S5-413
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Atrophic Vaginitis; Atrophy; Vaginitis
Keywords: Postmenopause; Vaginitis
MeSH Terms: conditions — Atrophic Vaginitis; Atrophy; Vaginitis | interventions — Polyvinyl Chloride

INTERVENTIONS:
Drug: PVC (daily for 21 days, 7 days off)
Drug: PVC (twice weekly)

SUMMARY:
This protocol is designed to study the effect and safety of 2 low-dose regimens of conjugated estrogen cream (PVC) given vaginally in postmenopausal women with atrophic vaginitis.

ELIGIBILITY:
Inclusion Criteria:

Generally healthy postmenopausal women with symptoms of atrophic vaginitis including vaginal dryness, vaginal itching, vaginal burning, and/or painful intercourse.

The subject must have a clinical diagnosis of atrophic vaginitis and an intact uterus.

Exclusion Criteria:

Women who do not have a clinical diagnosis of atrophic vaginitis.

Ages: 45 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 480
Dates: Start 2005-08; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of 2 low dose regimens of conjugated estrogen in the treatment of atrophic vaginitis from baseline to 12 weeks.

SECONDARY OUTCOMES:
To evaluate change from baseline in the percentage of superficial cells, symptom relief, the effect of both regimens on endometrial stimulation and genital health.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Principal Investigator — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (44):
- United States (31):
  - Tucson, Arizona
  - Encinitas, California
  - San Diego, California
  - Torrance, California
  - Aurora, Colorado
  - Brooksville, Florida
  - Miami, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Metairie, Louisiana
  - Troy, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - New Brunswick, New Jersey
  - Chapel Hill, North Carolina
  - Winston-Salem, North Carolina
  - Oklahoma City, Oklahoma
  - Danville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Carrollton, Texas
  - Colleyville, Texas
  - Dallas, Texas
  - Houston, Texas
  - Plano, Texas
  - Charlottesville, Virginia
  - Norfolk, Virginia
- Canada (13):
  - Calgary, Alberta
  - Coquitlam, British Columbia
  - Langley, British Columbia
  - Winnipeg, Manitoba
  - Kingston, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - MontrÃ©al, Quebec
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - QuÃ©bec, Quebec
  - Shawinigan, Quebec
  - Sherbrooke, Quebec